CLINICAL TRIAL: NCT00718042
Title: Evaluation of ABBOTT PRISM Chagas Assay and Chagas Confirmatory Assay
Brief Title: Evaluation of Chagas Blood Screening and Confirmatory Assays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diagnostics Division (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 7B5-02-06P06
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: healthy donors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): All subjects will have their blood tested by the investigational Chagas screening assay.
  Interventions: Device: ABBOTT PRISM Chagas Assay and Chagas Confirmatory Assay
- 2 (Experimental): Testing of blood donor samples with the investigational Chagas screening assay. Samples that test positive will be also tested with the Chagas confirmatory assay.
  Interventions: Device: ABBOTT PRISM Chagas Assay and Chagas Confirmatory Assay

INTERVENTIONS:
Device: ABBOTT PRISM Chagas Assay and Chagas Confirmatory Assay — Test blood donor sample with ABBOTT PRISM Chagas assay. If results are reactive, donor sample will be tested with Chagas Confirmatory assay. Donors reactive with screening assay or positive with confirmatory assay will be deferred and asked to return for a follow-up blood draw.
  Arms: 1
Device: ABBOTT PRISM Chagas Assay and Chagas Confirmatory Assay — Test blood donor sample with investigational Chagas assay. If results are reactive, donor samples will be tested with Chagas confirmatory assay. Donors reactive with screening assay or positive with confirmatory assay will be deferred and asked to return for a follow-up blood draw.
  Arms: 2

SUMMARY:
Protocol designed to test blood samples from blood donors of whole blood and blood components using a new investigational screening test (PRISM Chagas) that detects antibody to T. cruzi (Chagas infection). Results will be compared to the current T. cruzi antibody screening assay. Specimens positive with the screening assay will be further tested with a new investigational Chagas confirmatory assay [Enzyme Strip Assay (ESA) Chagas]. Additional specimens collected under separate protocols or sourced from suppliers will also be provided to the clinical sites for testing with PRISM Chagas assay and ESA Chagas.

ELIGIBILITY:
Inclusion Criteria:

* Healthy donors that have consented to participate in study

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41862 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Stramer, PhD, Principal Investigator — American National Red Cross; Sharon Gordon, Principal Investigator — Lifesource; Norman Kalmin, MD, Principal Investigator — South Texas Blood and Tissue Center; Carolyn T Young, MD, Principal Investigator — Rhode Island Blood Center; Deborah Williams, Principal Investigator — Florida Blood Services; Pauline Simmonds-Brown, Principal Investigator — Blood Net USA
Locations (7):
- United States (7):
  - BloodNet USA, Lakeland, Florida
  - Florida Blood Services, St. Petersburg, Florida
  - LifeSource Blood Center, Glenview, Illinois
  - American Red Cross Charlotte NTL, Charlotte, North Carolina
  - American Red Cross, Portland, Oregon
  - Rhode Island Blood Center, Providence, Rhode Island
  - South Texas Blood and Tissue Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: US blood donors specimens collected as part of routine blood donation (Specificity: 16313, Extended: 25549). Additional specimens included: 204 T cruzi antibody positive US blood donor; 110 parasite positive, 85 antibody positive, 525 Chagas endemic; and 330 unidentified US blood donor presumed T cruzi antibody negative were provided by Abbott.
Pre-assignment Details: All subjects were assigned to one group and tested with the PRISM Chagas assay. There were no pre-screening criteria.
  Specimens repeatedly reactive with the screening assay were further evaluated with ESA Chagas.
  The 330 unidentified US blood donor specimens presumed T cruzi antibody negative were only tested with ESA Chagas.
Groups:
- ABBOTT PRISM Chagas Specificity: All blood donor specimens tested by the investigational Chagas screening test in design validation phase.
- Reactivity T Cruzi Antibody Positive: Specimen antibody positive for T cruzi antibody collected in South America (85) under separate specimen collection protocols and unidentified US blood donor specimens (202) were tested with investigational Chagas screening assay and with the Chagas confirmatory assay.
- Reactivity in Chagas Endemic Population: Specimen collected in Chagas endemic area in South/Central America (524) under separate specimen collection protocol were tested with investigational Chagas screening assay and with the Chagas Confirmatory assay.
- Sensitivity Chagas Parasitology Positive Specimens: Specimen collected in South/Central America under separate specimen collection protocols were tested with investigational Chagas screening assay and with ESA Chagas.
- Chagas Extended Evaluation: US blood donor specimen were tested with investigational Chagas screening assay to identify repeatedly reactive specimens.
- ESA Chagas Specificity: US blood donor specimen presumed antibody negative for T cruzi antibody were tested with investigational ESA Chagas.
Period: ABBOTT PRISM Chagas Testing
Arm/Group | ABBOTT PRISM Chagas Specificity | Reactivity T Cruzi Antibody Positive | Reactivity in Chagas Endemic Population | Sensitivity Chagas Parasitology Positive Specimens | Chagas Extended Evaluation | ESA Chagas Specificity
Started | 16313 | 289 | 525 | 110 | 25549 | 0 (Specimens not screened with PRISM Chagas assay per protocol.)
Completed | 16249 | 287 | 524 | 110 | 25511 | 0
Not Completed | 64 | 2 | 1 | 0 | 38 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 64 | 0 | 0 | 0 | 36 | 0
Not completed — Insufficient sample | 0 | 1 | 1 | 0 | 0 | 0
Not completed — No result on comparator assay | 0 | 1 | 0 | 0 | 0 | 0
Period: ESA Chagas Testing
Arm/Group | ABBOTT PRISM Chagas Specificity | Reactivity T Cruzi Antibody Positive | Reactivity in Chagas Endemic Population | Sensitivity Chagas Parasitology Positive Specimens | Chagas Extended Evaluation | ESA Chagas Specificity
Started | 36 (Only specimens repeatedly reactive by screening assay or PRISM grayzone tested with ESA Chagas) | 287 | 524 | 110 | 43 (Only specimens repeatedly reactive by screening assay or PRISM grayzone tested with ESA Chagas) | 330 (Specimens only tested with ESA Chagas)
Completed | 36 | 287 | 524 | 110 | 43 | 330
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Donor Follow-up
Arm/Group | ABBOTT PRISM Chagas Specificity | Reactivity T Cruzi Antibody Positive | Reactivity in Chagas Endemic Population | Sensitivity Chagas Parasitology Positive Specimens | Chagas Extended Evaluation | ESA Chagas Specificity
Started | 36 | 0 (Follow-up not performed for this specimen population.) | 0 (Follow-up not performed for this specimen population.) | 0 (Follow-up not performed for this specimen population.) | 43 | 0 (Follow-up not performed for this specimen population.)
Completed | 23 | 0 | 0 | 0 | 24 | 0
Not Completed | 13 | 0 | 0 | 0 | 19 | 0
Not completed — Lost to Follow-up | 13 | 0 | 0 | 0 | 19 | 0

BASELINE CHARACTERISTICS:
Groups:
- ABBOTT PRISM Chagas Specificity; Chagas Extended Evaluation: All subject's blood tested by the investigational Chagas screening test.
- Total: Total of all reporting groups
Arm/Group | ABBOTT PRISM Chagas Specificity | Reactivity T Cruzi Antibody Positive | Reactivity in Chagas Endemic Population | ESA Chagas Specificity | Sensitivity Chagas Parasitology Positive Specimens | Chagas Extended Evaluation | Total
Number analyzed (Participants) | 16313 | 289 | 525 | 330 | 110 | 25549 | 43116
Age, Customized [Number; unit: Participants] — Age was not collected for this study.
  Participants
    >= 18 years | 16313 | 85 | 525 | 330 | 110 | 25549 | 42912
    Not Collected | 0 | 204 | 0 | 0 | 0 | 0 | 204
Sex/Gender, Customized [Number; unit: Participant] — Gender was not collected for all study populations.
  Participant
    Female | 0 | 44 | 336 | 0 | 53 | 0 | 433
    Male | 0 | 41 | 189 | 0 | 57 | 0 | 287
    Not Collected | 16313 | 204 | 0 | 330 | 0 | 25549 | 42396
Region of Enrollment [Number; unit: participants]
  United States | 16313 | 204 | 0 | 330 | 0 | 25549 | 42396
  Argentina | 0 | 85 | 176 | 0 | 76 | 0 | 337
  Brazil | 0 | 0 | 50 | 0 | 7 | 0 | 57
  Guatemala | 0 | 0 | 149 | 0 | 0 | 0 | 149
  Panama | 0 | 0 | 50 | 0 | 0 | 0 | 50
  Peru | 0 | 0 | 100 | 0 | 5 | 0 | 105
  Bolivia | 0 | 0 | 0 | 0 | 22 | 0 | 22

OUTCOME MEASURES:

1. Primary Outcome: PRISM Chagas Specificity
Description: Total of 16,249 serum and plasma blood donor specimens tested with PRISM Chagas assay during design validation phase. Repeatedly reactive specimens were tested further with a supplemental assay [radioimmune precipitation assay (RIPA)].
Time Frame: 6 months
Population: All fresh blood donor specimens tested with PRISM Chagas assay during design validation phase per protocol.
Measure: Number; unit: participants
Groups:
- ABBOTT PRISM Chagas Specificity: Specificity will be determined for the blood donor specimens tested with the investigational PRISM Chagas screening test.
Arm/Group | ABBOTT PRISM Chagas Specificity
Number analyzed (Participants) | 16249
participants
  PRISM Chagas Reactive, RIPA Negative | 23
  PRISM Chagas Nonreactive | 16223
  PRISM Chagas Reactive, RIPA Positive | 3
Statistical Analysis 1: Comparison: ABBOTT PRISM Chagas Specificity; Test type: Superiority or Other; Point Estimate; Specificity = 99.86, 95% CI 2-sided [99.79 to 99.91] — Numerator = All blood donors tested nonreactive from all True Negative blood donors (16,223) Denominator = All True Negative blood donors (16,246) True Negative excludes donor specimens positive by supplemental testing (3)

2. Secondary Outcome: PRISM Chagas Reactivity Serology Positive Specimens
Description: Total of 85 specimens from subjects from South America known to be positive for T cruzi antibodies and 202 US blood donor specimens that were repeatedly reactive on a licensed test for antibodies to T cruzi were tested with the PRISM Chagas assay and supplemental testing (RIPA).
Time Frame: 4 months
Population: Total of 287 specimens presumed T cruzi antibody positive per protocol.
Measure: Number; unit: participants
Groups:
- Reactivity T Cruzi Antibody Positive: Specimen positive for T cruzi antibody collected in South America (85) under separate specimen collection protocol and unidentified US blood donor specimens repeatedly reactive by T cruzi antibody licensed screening assay (202) were tested with investigational PRISM Chagas screening assay.
Arm/Group | Reactivity T Cruzi Antibody Positive
Number analyzed (Participants) | 287
participants
  PRISM Chagas Reactive, RIPA Positive | 224
  PRISM Chagas Reactive, RIPA Negative | 24
  PRISM Chagas Nonreactive, RIPA Negative | 39
  PRISM Chagas Nonreactive, RIPA Positive | 0

3. Primary Outcome: PRISM Chagas Sensitivity
Description: Specimens from subjects known to be T cruzi parasite positive were tested with PRISM Chagas assay.
Time Frame: 6 months
Population: Specimens from 110 individuals known to be positive for T cruzi parasite were tested with PRISM Chagas assay per protocol.
Measure: Number; unit: participants
Groups:
- Sensitivity Chagas Parasitology Positive Specimens: Specimen collected in South/Central America under separate specimen collection protocols were tested with investigational Chagas screening assay.
Arm/Group | Sensitivity Chagas Parasitology Positive Specimens
Number analyzed (Participants) | 110
participants
  PRISM Chagas Nonreactive | 0
  PRISM Chagas Reactive, Parasite Positive | 110
Statistical Analysis 1: Comparison: Sensitivity Chagas Parasitology Positive Specimens; Test type: Superiority or Other; Sensitivity; Point estimate = 100, 95% CI 2-sided [96.70 to 100.00]

4. Secondary Outcome: PRISM Chagas Reactivity in Chagas Endemic Population
Description: Population of specimen collected in Chagas endemic area in South/Central America (524) were tested to demonstrate reactivity with the PRISM Chagas assay in a population with a 5% or greater prevalence of infection with T cruzi antibody. specimens tested with PRISM Chagas assay and licensed test for T cruzi antibody and if repeatedly reactive with either assay the specimens were tested with supplemental assay (RIPA). Data presented with PRISM Chagas and RIPA results.
Time Frame: 2 months
Population: Total of 524 specimens from Chagas endemic areas tested with PRISM Chagas per protocol.
Measure: Number; unit: participants
Groups:
- PRISM Chagas Reactivity Endemic Population: Specimen collected in Chagas endemic area in South/Central America (524) under separate specimen collection protocol were tested with investigational Chagas screening assay and with the Chagas Confirmatory assay.
Arm/Group | PRISM Chagas Reactivity Endemic Population
Number analyzed (Participants) | 524
participants
  PRISM Chagas Reactive, RIPA Positive | 129
  PRISM Chagas Reactive, RIPA Negative | 5
  PRISM Chagas Reactive, RIPA Indeterminate | 3
  PRISM Chagas Nonreactive, RIPA Positive | 2
  PRISM Chagas Nonreactive, RIPA Negative | 385
  PRISM Chagas Nonreactive, RIPA Indeterminate | 0

5. Secondary Outcome: ESA Chagas Testing of US Blood Donor Specimens Repeatedly Reactive by ABBOTT PRISM Chagas.
Description: A total of 41,760 US blood donor specimens were tested by ABBOTT PRISM Chagas. Of these specimens, 58 out of 79 specimens were T cruzi antibody repeatedly reactive by ABBOTT PRISM Chagas (26 from 16,249 donor specimens tested in design validation phase and 32 from 25,511 specimens from the Chagas extended evaluation). Donor specimens that were repeatedly reactive with the licensed T cruzi antibody assay, but PRISM Chagas nonreactive (6) and specimens PRISM Chagas grayzone negative (15) were excluded from this analysis.
Time Frame: 15 months
Population: A total of 58 US blood donor specimens were PRISM Chagas repeatedly reactive were included per protocol.
Measure: Number; unit: participants
Groups:
- ESA Chagas US Donor Specimen Testing: A total of 58 PRISM Chagas repeatedly reactive US blood donor specimens tested with both ESA Chagas and RIPA.
Arm/Group | ESA Chagas US Donor Specimen Testing
Number analyzed (Participants) | 58
participants
  ESA Chagas Positive, RIPA Positive | 9
  ESA Chagas Positive, RIPA Negative | 49

6. Primary Outcome: ESA Chagas Specificity
Description: Preselected US blood donor specimens (330) presumed T cruzi antibody negative negative that were tested only with the investigational ESA Chagas.
Time Frame: 3 months
Population: Determine percentage of donor specimens ESA Chagas negative in a presumed negative population per protocol.
Measure: Number; unit: participants
Arm/Group | ESA Chagas Specificity
Number analyzed (Participants) | 330
participants
  ESA Chagas Negative | 327
  ESA Chagas Indeterminate | 3
  ESA Chagas Positive | 0
Statistical Analysis 1: Comparison: ESA Chagas Specificity; Test type: Superiority or Other; Percentage Negative; Percentage = 99.1, 95% CI 2-sided [97.4 to 99.8]

7. Primary Outcome: ESA Chagas Sensitivity
Description: Specimens from individuals known to be T cruzi parasite positive were tested with ESA Chagas assay.
Time Frame: 3 months
Population: Specimens from 110 subjects known to be positive for T cruzi parasite tested with ESA Chagas per protocol.
Measure: Number; unit: participants
Groups:
- Sensitivity Chagas Parasitology Positive Specimens: Specimen collected in South or Central America under separate specimen collection protocols were tested with investigational with ESA Chagas.
Arm/Group | Sensitivity Chagas Parasitology Positive Specimens
Number analyzed (Participants) | 110
participants
  ESA Chagas Positive | 110
  ESA Chagas Negative | 0

8. Secondary Outcome: ESA Chagas Sensitivity in Serologically Positive Non-US Specimens
Description: ESA Chagas Sensitivity in a non-US population was determined for the 85 out of the total 287 serologically positive specimens (202 US Serology Positive specimens were excluded). These specimens were collected from individuals positive for T cruzi antibodies based on 2 different serologic tests for antibodies to T cruzi in Argentina and were tested with ESA Chagas.
Time Frame: 3 months
Population: A total of 85 serum specimens from non-US individuals reactive for T cruzi antibodies per protocol.
Measure: Number; unit: participants
Groups:
- ESA Chagas Non-US Serologically Positive: Specimen antibody positive for T cruzi antibody collected in South America (85) under separate specimen collection protocols.
Arm/Group | ESA Chagas Non-US Serologically Positive
Number analyzed (Participants) | 85
participants
  ESA Chagas Positve | 85
  ESA Chagas Negative | 0

9. Secondary Outcome: ESA Chagas Testing in Chagas Endemic Population
Description: Specimen collected in Chagas endemic areas in South or Central America (524) tested with ESA Chagas and licensed test for T cruzi antibody. Specimens repeatedly reactive with either screening assay and/or ESA Chagas positive were tested with supplemental assay (RIPA). Presentation of ESA Chagas results for 132 specimens from a Chagas endemic population that were RIPA positive.
Time Frame: 2 months
Population: Total of 132 out of the 524 specimens from Chagas endemic areas that were tested RIPA positive per protocol.
Measure: Number; unit: participants
Groups:
- Reactivity in Chagas Endemic Population: Specimen from Chagas endemic area in South or Central America (524) under separate specimen collection protocol were tested with investigational ESA Chagas.
Arm/Group | Reactivity in Chagas Endemic Population
Number analyzed (Participants) | 132
participants
  ESA Chagas Postive, RIPA Positive | 130
  ESA Chagas Indeterminate, RIPA Positive | 2

ADVERSE EVENTS:
Time Frame: Adverse event data collected during donor follow-up collection for period of 10 months. Donors reactive with screening assay or positive with confirmatory assay will be deferred and asked to return for a follow-up blood draw.
Description: Adverse events were not applicable for blood donor specimens tested that were collected as part of routine blood donation and specimens provided by Abbott to testing sites.
Groups:
- Donor Follow-up Specimen Collection: Blood donors
Arm/Group | Donor Follow-up Specimen Collection
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must provide a copy of any proposed publication/presentation at least 30 days prior to submission for sponsor's review/approval. The PI must incorporate changes as the sponsor requires in order to protect the sponsor's proprietary rights and interests. The sponsor may require the PI to include acknowledgement of the sponsor's role in the study. The PI may be requested to delay publication/presentation an extra 60 days to enable sponsor to secure patent or other proprietary protection.